CLINICAL TRIAL: NCT04487522
Title: RECOVER: a PRospECtive EvaluatiOn of Pain After Retromuscular VEntRal Hernia Repair
Brief Title: Pain and Quality of Life After Retromuscular Ventral Hernia Repair (RECOVER)
Acronym: RECOVER
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: RECOVER
Record Dates: First submitted 2020-07-08; First posted 2020-07-27 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retromuscular ventral hernia repair: These subjects will undergo an open, a laparoscopic, or a robotic-assisted retromuscular ventral hernia repair.
  Interventions: Procedure: Open retromuscular ventral hernia repair; Procedure: Laparoscopic retromuscular ventral hernia repair; Device: Robotic-assisted retromuscular ventral hernia repair
- Retromuscular TAR ventral hernia repair: These subjects will undergo an open or a robotic-assisted retromuscular transversus abdominis release (TAR) ventral hernia repair.
  Interventions: Procedure: Open retromuscular ventral hernia repair; Device: Robotic-assisted retromuscular ventral hernia repair

INTERVENTIONS:
Procedure: Open retromuscular ventral hernia repair — With the subject under general anesthesia, a single incision is made in the abdomen. The retrorectus space is developed for mesh placement to repair the defect. The repair technique will be per the surgeon's standard of care.
Procedure: Laparoscopic retromuscular ventral hernia repair — With the subject under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and laparoscopic instruments as well as a laparoscope are inserted to complete the repair. The retrorectus space is developed for mesh placement to repair the defect. The repair technique will be per the surgeon's standard of care.
  Groups: Retromuscular ventral hernia repair
Device: Robotic-assisted retromuscular ventral hernia repair — With the patient under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and the da Vinci Robotic Surgical System (Intuitive) is docked to the subject and used to complete the procedure. The retrorectus space is developed for mesh placement to repair the defect. The repair technique will be per the surgeon's standard of care.

SUMMARY:
The study aims to explore the difference in outcomes relating to pain and quality of life after open, laparoscopic, and robotic-assisted retromuscular ventral hernia repair.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational study assessing outcomes relating to pain and quality of life for subjects undergoing open, laparoscopic, or robotic-assisted retromuscular ventral hernia repair. The study will focus on short-term post-operative outcomes through 3 months. The study will also collect recurrence data through 1 year. During the post-operative period through 3 months, pain medication intake, subject reported pain (on post-operative day 7, 14, 21, 28, and 3 months) and quality of life (on day 28, 3 months, and 1 year) and incidence of intra-operative and post-operative adverse events related to the ventral hernia repair will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 89 years of age
* Subject is a candidate for an elective retromuscular ventral hernia repair under general anesthesia
* Subject has access to complete study assessments electronically and agrees to comply with all follow-up requirements
* Ventral hernia is >= 4cm

Exclusion Criteria:

* Subject who will have an emergent hernia repair
* Subject has a parastomal hernia (i.e. hernia related to ostomy formation)
* Subject with a history of chronic pain and/or taking daily pain medication for >6 weeks
* Subject wtih a history of substance abuse (excluding marijuana) and/or current (within 30 days) narcotic use
* Subject with a history of MRSA infection
* Subject with HbA1c level > 8.5%
* Subject undergoing a minimally invasive (MIS) repair who will require the use of Exparel during the surgical procedure
* Subject who will undergo a concomitant hernia repair or any other concomitant procedure
* Subject has cirrhosis
* Current nicotine use (including vaping) within the past 30 days
* Subject is contraindicated for general anesthesia or surgery
* Subject has a known bleeding or clotting disorder
* Pregnant or suspected pregnancy
* Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with the study requirements or ability to provide informed consent
* Subject belonging to other vulnerable population, e.g., prisoner or ward of state
* Subject is currently participating in another interventional research study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who will undergo an elective retromuscular ventral hernia repair procedure and who meet all eligibility criteria will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Pain scores | 7 days
  Subject reported pain scores assessed by the Subject-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey.
Narcotic usage | 4 weeks
  Narcotic usage (in hospital and out of hospital) taken for the purpose of managing abdominal pain after the ventral hernia repair.
Non-opioid prescription pain medication usage | 4 weeks
  Non-opioid prescription pain medication usage related to the retromuscular ventral hernia repair

SECONDARY OUTCOMES:
Narcotic usage | 3 months
  Narcotic usage related to the retromuscular ventral hernia repair.
Non-opioid prescription pain medication usage | 3 months
  Non-opioid prescription pain medication usage related to the retromuscular ventral hernia repair.
Over the counter pain medication usage | 4 weeks
  Over the counter (OTC) pain medication usage after the retromuscular ventral hernia repair procedure as determined by patient reporting of OTC pain medication usage at follow-ups
Need for refill prescription pain medication | 4 weeks
  Need for refill of prescription pain medication after the retromuscular ventral hernia repair
PROMIS 3a pain scores | 4 weeks
  Subject reported pain scores assessed by the Subject-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey.
Hospital length of stay | Start of procedure to discharge from the hospital (check out time), up to an approximate of one week
  Duration of hospital stay
Incidence of intraoperative adverse events related to the retromuscular ventral hernia repair | intraoperatve
  Intra-operative adverse events related to the retromuscular ventral hernia repair
Incidence of postoperative adverse events related to the retromuscular ventral hernia repair | 3 months
  Post-operative adverse events related to the retromuscular ventral hernia repair
Hernia recurrence | 1 year
  Hernia recurrence after the retromuscular ventral hernia repair
EQ-5D-3L QOL scores | 4 weeks
  Quality of life assessment using the EQ-5D-3L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kaiser Foundation Research Institute, Oakland/Richmond, Oakland, California
  - Kaiser Foundation Research Institute, South Sacramento, Sacramento, California
  - Kaiser Foundation Research Institute, Santa Clara, Santa Clara, California
  - Kaiser Foundation Research Institute, Walnut Creek, Walnut Creek, California